CLINICAL TRIAL: NCT00113295
Title: Combination of Paroxetine CR and Quetiapine for the Treatment of Refractory Generalized Anxiety Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Naomi M. Simon, Director, Center for Anxiety and Traumatic Stress Disorders, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2003-P001805
Record Dates: First submitted 2005-06-07; First posted 2005-06-08 (Estimated); Results first posted 2014-04-23 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-03

CONDITIONS: Anxiety Disorder
Keywords: generalized anxiety disorder; pharmacotherapy; treatment refractory; double-blind
MeSH Terms: conditions — Anxiety Disorders; Generalized Anxiety Disorder | interventions — Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Paroxetine CR and Placebo (Active Comparator): Eleven individuals were randomized to plaecbo augmentation of continued paroxetine CR at the week 10 dose level. In the first phase of the study, individuals started at 12.5 mg/day of paroxetine and flexibly titrated up to a maximum of 62.5 mg/day by week 10. Individuals who did not achieve remission and were randomized into the placebo group received placebo augmentation of continued paroxetine CR at the week 10 dose level.
  Interventions: Drug: Continued Paroxetine CR; Drug: Placebo
- Quetiapine and continued paroxetine CR (Experimental): Eleven individuals were randomized to quetiapine augmentation of continued paroxetine CR at the week 10 dose level. In the first phase of the study, individuals started at 12.5 mg/day of paroxetine and flexibly tirated up to a maximum of 62.5 mg/day by week 10. Individuals who did not receive remission and were randomized to receive quetiapine started at 25 mg at bedtime for the first week, then flexibly dosed based on response and tolerability to a maximum of 200 mg BID by week 16.
  Interventions: Drug: Continued Paroxetine CR; Drug: Quetiapine

INTERVENTIONS:
Drug: Continued Paroxetine CR
Drug: Quetiapine
  Arms: Quetiapine and continued paroxetine CR
Drug: Placebo
  Arms: Paroxetine CR and Placebo

SUMMARY:
The purpose of this study is to examine the safety and efficacy of quetiapine for generalized anxiety disorder patients who remain symptomatic despite treatment with paroxetine CR.

DETAILED DESCRIPTION:
Generalized anxiety disorder (GAD) is a relatively common condition affecting 5% of the population, with a typically chronic course and associated with significant psychosocial impairment and decreased quality of life (Schweizer, 1995). Although a number of therapeutic agents demonstrate some efficacy in the treatment of generalized anxiety disorder, only a minority of anxious patients experience remission with initial treatment.

The purpose of this study is to examine the efficacy of one strategy, the addition of quetiapine, for the treatment of patients with GAD who remain refractory despite an adequate treatment trial with a selective serotonin reuptake inhibitor (SSRI). This is an investigator-initiated augmentation study of an already approved drug for a different indication. Quetiapine is a novel antipsychotic agent with potent effects at the serotonergic, as well as dopaminergic receptor, and a more favorable side effect profile than standard neuroleptics, including a low potential to cause extrapyramidal symptoms.

This is a two phase, 18-week research study in which participants who remain symptomatic at the end of one phase (10 weeks) enter into the next phase. In phase I, all participants receive paroxetine CR (Paxil CR) for 10 weeks. Participants who continue to have anxiety symptoms will enter the 8-week Phase II, in which they continue taking Paxil CR and they will also be randomly assigned (by chance, like a flip of a coin) to receive quetiapine (Seroquel) or placebo (contains no active medication).

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients, age 18-72.
* Primary diagnosis of generalized anxiety disorder.
* Patients on concurrent benzodiazepines will be entered into the trial if they remain symptomatic despite stable doses for at least one month

Exclusion Criteria:

* Pregnant or lactating women or other women of child bearing potential not using acceptable means of birth control
* Patients with a primary diagnosis of major depression, dysthymia, panic disorder or social phobia.
* Patients with current or history of bipolar disorder, schizophrenia or other psychotic conditions
* Patients with post-traumatic stress disorder or obsessive-compulsive disorder current in the past 6 months.
* Patients with a history of alcohol or substance abuse or dependence within the last six months.
* Patients with significant unstable medical illness.
* Ongoing psychotherapy directed toward the treatment of generalized anxiety disorder.
* History of hypersensitivity to paroxetine CR, paroxetine or quetiapine.
* History of cataracts.
* Concurrent use of psychotropic medications including buspirone and antidepressants. Patients must have discontinued buspirone or antidepressant therapy at least two weeks prior to study entry, and fluoxetine at least four weeks prior, but no patient will be taken off effective medication.
* Concomitant use of herbs and dietary supplements with known psychotropic properties, including St John's Wort, Kava, Valerian, Gingko, Ginseng, ephedra and weight loss supplements. Other than such agents with known psychotropic properties, no over the counter medications are exclusionary.

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2004-02; Primary Completion 2007-02 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naomi M Simon, MD, Principal Investigator — Massachusetts General Hospital; Kathryn Connors, MD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Duke University Medical Center, Durham, North Carolina

REFERENCES:
- See also: The Center for Anxiety and Traumatic Stress Disorders at Massachusetts General Hospital — http://www.mghanxiety.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One hundred and one individuals were recruited through advertisement and clinical referral from February 2004 to June 2007, signed consent, and participated in a screening visit. Fifty-four individuals (53.5%) with GAD met the study entry criteria and initiated paroxetine CR in phase 1 of the trial.
Pre-assignment Details: Seven patients did not complete phase 1. Of phase 1 completers, 21 were not randomized. Twenty-two patients were randomized, 11 to quetiapine and 11 to placebo augmentation.
  *Note that the data reported throughout the results section are from Phase 2 only.
Groups:
- Quetiapine, 25-400mg/Day Augmentation of Continued Paroxetine: In the first phase of the study, individuals started at 12.5 mg/day of paroxetine and flexibly tirated up to a maximum of 62.5 mg/day by week 10. Individuals who did not receive remission and were randomized to receive quetiapine started at 25 mg at bedtime for the first week, then flexibly dosed based on response and tolerability to a maximum of 200 mg BID by week 16.
- Placebo Augmentation of Continued Paroxetine: In the first phase of the study, individuals started at 12.5 mg/day of paroxetine and flexibly titrated up to a maximum of 62.5 mg/day by week 10. Individuals who did not achieve remission and were randomized into the placebo group received placebo augmentation of continued paroxetine CR at the week 10 dose level.
Period: Overall Study
Arm/Group | Quetiapine, 25-400mg/Day Augmentation of Continued Paroxetine | Placebo Augmentation of Continued Paroxetine
Started | 11 | 11
Completed | 6 | 10
Not Completed | 5 | 1
Not completed — Adverse Event | 4 | 1
Not completed — Unrelated Medical Illness | 1 | 0

BASELINE CHARACTERISTICS:
Population: Eligible participants were men or women aged 18 and older with a primary diagnosis of DSM-IV GAD.
Groups:
- Quetiapine, 25-400mg/Day Augmentation of Continued Paroxetine: Individuals randomized to receive Quetiapine started at 25 mg at bedtime for the first week, then flexibly dosed based on response and tolerability to a maximum of 200 mg BID by week 16.
- Placebo Augmentation of Continued Paroxetine: Individuals received placebo augmentation of continued paroxetine CR at the week 10 dose level.
- Total: Total of all reporting groups
Arm/Group | Quetiapine, 25-400mg/Day Augmentation of Continued Paroxetine | Placebo Augmentation of Continued Paroxetine | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Continuous [Mean (Standard Deviation); unit: years]
  At Phase 2 Baseline | 43.8 (12.5) | 40.5 (11.2) | 42.2 (11.7)
Sex/Gender, Customized [Number; unit: participants]
  Phase 2 Baseline Females | 4 | 7 | 11
  Phase 2 Baseline Males | 7 | 4 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 10 | 8 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
HAM-A [Mean (Standard Deviation); unit: units on a scale] — The 14-item Hamilton Anxiety Rating Scale (HAM-A) (Hamilton, 1959) was developed to assess anxiety in a clinical population. It is considered a measure of general anxiety across anxiety disorders, in addition to being a gold standard measure for GAD.
  units on a scale | 16.27 (5.04) | 15.82 (4.77) | 16.05 (4.8)
CGI-S [Mean (Standard Deviation); unit: Units on a scale] — The Clinical Global Impression of Improvement (CGI-I) measures illness severity and improvement. The patient's current condition is compared to the patient's baseline condition on a seven-point scale. The condition is rated as 1=very much improved since the initiation of treatment; 2=much improved; 3=minimally improved; 4=no change from baseline (the initiation of treatment); 5=minimally worse; 6= much worse; 7=very much worse since the initiation of treatment.
  Units on a scale | 3.64 (0.67) | 3.91 (0.83) | 3.77 (0.75)
MADRS [Mean (Standard Deviation); unit: units on a scale] — The Montgomery-Asberg Depression Rating Scale (MADRS) measures depressive symptoms.
  units on a scale | 11.45 (1.93) | 12.36 (4.80) | 11.91 (3.66)
Q-LES-Q [Mean (Standard Deviation); unit: units on a scale] — The Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) measures the degree of enjoyment and satisfaction experienced by subjects in various areas of daily functioning.
  units on a scale | 45.13 (10.6) | 45.89 (8.88) | 45.51 (9.77)

OUTCOME MEASURES:

1. Secondary Outcome: Remission (HAM-A ≤ 7)
Description: Remission was measured as a secondary outcome using a score of less than or equal to 7 on the Hamilton Anxiety Scale (HAM-A).
Time Frame: Week 18 (Study Endpoint)
Measure: Number; unit: participants
Arm/Group | Quetiapine, 25-400mg/Day Augmentation of Continued Paroxetine | Placebo Augmentation of Continued Paroxetine
Number analyzed (Participants) | 11 | 11
participants | 4 | 2

2. Primary Outcome: Hamilton Anxiety Scale (HAM-A) Score at Study Endpoint.
Description: Symptoms of generalized anxiety disorder as measured by the Hamilton Anxiety Scale (HAM-A) at week 18/study endpoint. Each item is scored on a scale from 0 (not present) to 4 (severe) with a total score range of 0-56. Changes in HAM-A scores are calculated as the difference between the baseline HAM-A scores and scores at week 18/study endpoint.
  The 14-item Hamilton Anxiety Rating Scale (HAM-A) (Hamilton, 1959) was developed to assess anxiety in a clinical population. It is considered a measure of general anxiety across anxiety disorders, in addition to being a gold standard measure for GAD.
Time Frame: Baseline and Week 18
Population: Twenty-two patients were randomized, 11 to quetiapine and 11 to placebo augmentation, and all had at least one assessment postrandomization and were included in the phase 2 efficacy analyses; of this group, six randomized to quetiapine (54.5%) and ten to placebo (90.1%) completed the trial.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Quetiapine, 25-400mg/Day Augmentation of Continued Paroxetine: Individuals randomized to receive Quetiapine started at 25 mg at bedtime for the first week, then flexibly dosed based on response and tolerability to a maximum of 200 mg BID by week 16(mean±SD endpoint dose=120.5±100.5 mg/day).
Arm/Group | Quetiapine, 25-400mg/Day Augmentation of Continued Paroxetine | Placebo Augmentation of Continued Paroxetine
Number analyzed (Participants) | 11 | 11
units on a scale
  Baseline | 16.27 (5.04) | 15.82 (4.77)
  Week 18 | 13.64 (8.36) | 15.55 (7.97)
  Change | -2.6 (5.8) | -0.3 (5.5)
Statistical Analysis 1: Comparison: Quetiapine, 25-400mg/Day Augmentation of Continued Paroxetine vs Placebo Augmentation of Continued Paroxetine; In phase 2, comprising randomized double-blind quetiapine augmentation, change scores were examined with two-tailed, two-sample t tests, utilizing scores at phase 2 randomization as baseline. All analyses were intention to treat (ITT) with the last visit carried forward (LVCF) for subjects that did not complete the study; Test type: Superiority or Other; p < 0.05, t-test, 2 sided — No adjustment for multiple testing; Mean Difference (Net) = 2.3 — This analysis applies to the additional reduction from phase 2 randomization to phase 2 endpoint in HAM-A scores

3. Secondary Outcome: Response, Clinical Global Impression of Improvement (CGI-I)
Description: Response was measured as a secondary outcome using the Clinical Global Impression of Improvement (CGI-I). Response was defined as a score of 1 ["very much improved"] or 2 ["much improved"] at study endpoint.
Time Frame: Week 18 (Phase 2 Endpoint)
Measure: Number; unit: participants
Arm/Group | Quetiapine, 25-400mg/Day Augmentation of Continued Paroxetine | Placebo Augmentation of Continued Paroxetine
Number analyzed (Participants) | 11 | 11
participants | 6 (0.8) | 5 (0.8)

4. Secondary Outcome: Depressive Symptoms, Montgomery-Asberg Depression Rating Scale (MADRS)
Description: Depressive symptoms were measured at a secondary outcome using the Montgomery-Asberg Depression Rating Scale (MADRS). Each item is scored on a scale of 1-6; The total score range is 0-60, with higher scores indicated higher levels of depression severity.
Time Frame: Week 10 (Phase 1 Endpoint) and Week 18 (Phase 2 Endpoint)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Quetiapine, 25-400mg/Day Augmentation of Continued Paroxetine | Placebo Augmentation of Continued Paroxetine
Number analyzed (Participants) | 11 | 11
units on a scale
  Baseline (Week 10) | 11.45 (1.93) | 12.36 (4.80)
  Endpoint (Week 18) | 10.27 (7.30) | 11.64 (5.92)

5. Secondary Outcome: The Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q).
Description: The 16-item Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) is used to assess quality of life changes with treatment. Total scores range from 14-70, with higher levels of satisfaction yielding higher scores.
Time Frame: Week 10 (Phase 1 Endpoint) and Week 18 (Phase 2 Endpoint)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Quetiapine, 25-400mg/Day Augmentation of Continued Paroxetine | Placebo Augmentation of Continued Paroxetine
Number analyzed (Participants) | 11 | 11
units on a scale
  Baseline (Week 10) | 45.13 (10.64) | 45.89 (8.88)
  Endpoint (Week 18) | 46.25 (9.45) | 45.11 (10.55)

ADVERSE EVENTS:
Time Frame: Adverse Event data was collected throughout the 18 week study period, both during Phase 1 (ten weeks) and Phase 2 (eight weeks).
Description: Safety evaluation included assessment of vital signs and weight at each visit and open-ended query regarding adverse events. The Simpson-Angus Scale (Simpson and Angus 1970) and the Barnes Akathisia Scale (Barnes 1989) were employed to assess for the development of akathisia and extrapyramidal side effects.
Groups:
- Paroxetine: Individuals received paroxetine CR for 10 weeks in Phase 1 of the study, initiated at 12.5 mg and flexibly titrated up to a maximum of 62.5 mg/day by week 8.
Arm/Group | Quetiapine, 25-400mg/Day Augmentation of Continued Paroxetine | Placebo Augmentation of Continued Paroxetine | Paroxetine
Serious Adverse Events (participants affected / at risk) | 2/11 | 1/11 | 0/50
Other Adverse Events (participants affected / at risk) | 7/11 | 8/11 | 6/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quetiapine, 25-400mg/Day Augmentation of Continued Paroxetine (N=11) | Placebo Augmentation of Continued Paroxetine (N=11) | Paroxetine (N=50)
Migraine Headache (General disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea and high fever (General disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Quetiapine, 25-400mg/Day Augmentation of Continued Paroxetine (N=11) | Placebo Augmentation of Continued Paroxetine (N=11) | Paroxetine (N=50)
Appetite Decrease (Metabolism and nutrition disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 2 | 1
Diarrhea (Gastrointestinal disorders) | 3 | 2 | 0
Dry mouth (General disorders) | 3 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 5
Headaches (General disorders) | 1 | 1 | 1
Insomnia (General disorders) | 1 | 3 | 0
Jittery/shaky/restless (General disorders) | 1 | 0 | 0
Nausea (General disorders) | 1 | 0 | 0
Sedation (General disorders) | 6 | 1 | 0
Sexual dysfunction (General disorders) | 2 | 3 | 0
Trouble Sleeping (General disorders) | 1 | 0 | 1
Urinary hesitancy (Renal and urinary disorders) | 1 | 0 | 0
Vivid Dreams (General disorders) | 1 | 3 | 0
Weight gain (Metabolism and nutrition disorders) | 0 | 2 | 0
Akathisia (General disorders) | 1 | 0 | 0
Difficulty Concentrating (General disorders) | 1 | 1 | 0
Forgetfulness (General disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 0
Gas (Gastrointestinal disorders) | 1 | 0 | 0
Irritability (General disorders) | 1 | 0 | 0
Myoclonic Jerks (General disorders) | 1 | 0 | 0
Morning Grogginess (General disorders) | 1 | 0 | 0
Spasm (General disorders) | 1 | 1 | 0
Appetite Increase (General disorders) | 1 | 0 | 0
Tremor (General disorders) | 1 | 0 | 0
Increased Sleep (General disorders) | 0 | 1 | 0
Sweating (General disorders) | 0 | 2 | 0

LIMITATIONS AND CAVEATS:
Relatively small sample size of the randomized controlled phase (phase 2); conclusions from the study are limited to low power; improvement in Phase I open label paroxetine CR may include "placebo" response to ancillary aspects of a treatment study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No